CLINICAL TRIAL: NCT01268098
Title: A Randomized, Dose-blinded Study to Investigate the Safety and Efficacy of NPSP558, a Recombinant Human Parathyroid Hormone [rhPTH(1-84)], at Fixed Doses of 25 µg and 50 µg for the Treatment of Adults With Hypoparathyroidism
Brief Title: Study of Safety and Efficacy of a rhPTH[1-84] of Fixed Doses of 25 and 50 mcg in Adults With Hypoparathyroidism (RELAY)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAR-C10-007
Record Dates: First submitted 2010-12-28; First posted 2010-12-29 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Hypoparathyroidism
Keywords: Hypoparathyroidism, rhPTH[1-84], NPSP558
MeSH Terms: conditions — Hypoparathyroidism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 25 µg dose (Experimental): 25 µg
  Interventions: Drug: NPSP558
- 50 µg dose (Experimental): 50 µg
  Interventions: Drug: NPSP558

INTERVENTIONS:
Drug: NPSP558 — All patients will inject NPSP558 25 or 50 µg SC QD into alternating thighs in the morning via a multidose injection pen device.
  Other Names: RELAY

SUMMARY:
Use of PTH (1-84) a recombinant hormone in 25 µg or 50 µg doses for the treatment of adults with hypoparathyroidism. The use of PTH (1-84) should result in a decrease of calcium and vitamin D supplements.

DETAILED DESCRIPTION:
Patients with a history of Hypoparathyroidism will be randomized to receive study drug for 8 weeks, which will be injected daily in either thigh. During that time they will be monitored for safety (specifically calcium levels in blood or urine). In addition, the patients' intake of Vitamin D and Calcium will be measured.

ELIGIBILITY:
Main Inclusion Criteria:

1. Previously completed 24 weeks of therapy and 4 weeks of follow-up in the REPLACE study
2. With regard to female patients: women who are postmenopausal or willing to use two medically acceptable methods of contraception for the duration of the study with pregnancy testing conducted at every scheduled office visit
3. Total serum calcium ≤ ULN based on local laboratory results prior to randomization
4. Serum 25(OH) vitamin D ≤ 1.5 times the ULN within approximately 8 weeks prior to randomization

Main Exclusion Criteria:

1. Any disease or condition that, in the opinion of the investigator, has a high probability of precluding the patient from completing the study or being able to appropriately comply with study requirements
2. Use of raloxifene hydrochloride or intravenous (IV) bisphosphonates since the end of participation in the REPLACE trial
3. Chronic (ie, ≥ 1 month exposure) use of systemic corticosteroids, oral bisphosphonates, calcitonin, fluoride tablets, or cinacalcet hydrochloride
4. Pregnant or lactating women
5. Any condition that would, in the investigator's opinion in consultation with the sponsor, preclude the safe use of PTH
6. Use of any experimental drug other than NPSP558 within 3 months of baseline.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-02-09 (Actual); Primary Completion 2011-09-23 (Actual); Study Completion 2011-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (12):
- United States (12):
  - Advance Medical Research LLC, Lakewood, California
  - University of Chicago Medical Center, Chicago, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan Bone & Mineral Clinic PC, Detroit, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Medical Center, New York, New York
  - University Physicians Group, Staten Island, New York
  - Physician East PA, Greenville, North Carolina
  - University of Cincinnati Bone Health and Osteoporosis Center, Cincinnati, Ohio
  - Cetero Research DGD Research Inc., San Antonio, Texas
  - The Vancouver Clinic, Vancouver, Washington

REFERENCES:
- [Derived] Ayodele O, Rejnmark L, Mu F, Lax A, Berman R, Swallow E, Gosmanova EO. Five-Year Estimated Glomerular Filtration Rate in Adults with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Nov;39(11):5013-5024. doi: 10.1007/s12325-022-02292-1. Epub 2022 Aug 26. PMID 36018496
- [Derived] Rejnmark L, Ayodele O, Lax A, Mu F, Swallow E, Gosmanova EO. The risk of chronic kidney disease development in adult patients with chronic hypoparathyroidism treated with rhPTH(1-84): A retrospective cohort study. Clin Endocrinol (Oxf). 2023 Apr;98(4):496-504. doi: 10.1111/cen.14813. Epub 2022 Aug 28. PMID 35974422
- [Derived] Ayodele O, Mu F, Berman R, Swallow E, Rejnmark L, Gosmanova EO, Kaul S. Lower Risk of Cardiovascular Events in Adult Patients with Chronic Hypoparathyroidism Treated with rhPTH(1-84): A Retrospective Cohort Study. Adv Ther. 2022 Aug;39(8):3845-3856. doi: 10.1007/s12325-022-02198-y. Epub 2022 Jun 11. PMID 35696069
- [Derived] Chen KS, Gosmanova EO, Curhan GC, Ketteler M, Rubin M, Swallow E, Zhao J, Wang J, Sherry N, Krasner A, Bilezikian JP. Five-year Estimated Glomerular Filtration Rate in Patients With Hypoparathyroidism Treated With and Without rhPTH(1-84). J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3557-65. doi: 10.1210/clinem/dgaa490. PMID 32738041
- [Derived] Bilezikian JP, Clarke BL, Mannstadt M, Rothman J, Vokes T, Lee HM, Krasner A. Safety and Efficacy of Recombinant Human Parathyroid Hormone in Adults With Hypoparathyroidism Randomly Assigned to Receive Fixed 25-mug or 50-mug Daily Doses. Clin Ther. 2017 Oct;39(10):2096-2102. doi: 10.1016/j.clinthera.2017.08.011. Epub 2017 Sep 21. PMID 28942334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 42 Subjects enrolled between 2/2011 and 9/2011 at 11 sites in the US.
Pre-assignment Details: Subjects who completed 24 wks of treatment and 4 wks follow-up in the REPLACE Study (NCT00732615) or received 2 single doses in Phase I Study C09-002 followed by a 4-wk washout, or enrolled in the REPLACE Study and entered into the optimization phase, but were not randomized due to the close of randomization; or were new to the NPSP558 program.
Groups:
- NPSP558 - 25 µg Dose: NPSP558: Recombinant Human Parathyroid hormone (rhPTH[1-84]) 25 mcg subcutaneously daily.
- NPSP558 - 50 µg Dose: NPSP558: Recombinant Human Parathyroid hormone (rhPTH[1-84]) 50 mcg subcutaneously daily.
Period: Overall Study
Arm/Group | NPSP558 - 25 µg Dose | NPSP558 - 50 µg Dose
Started | 19 | 23
Completed | 18 | 23
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NPSP558 - 25 µg Dose | NPSP558 - 50 µg Dose | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Customized [Count of Participants; unit: Participants]
  < 45 years | 6 | 8 | 14
  45 to 64 years | 10 | 15 | 25
  >/= 65 years | 3 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 3 | 4 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 17 | 22 | 39
  Asian | 1 | 1 | 2
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved the Primary Triple Endpoint at Week 8, Based on Investigator Prescribed Data.
Description: The triple efficacy endpoint criteria were defined as a reduction from baseline in oral calcium to ≤ 500 mg/day, a reduction from baseline in calcitriol dose to ≤ 0.25 µg/day, and an albumin-corrected total serum calcium level between 7.5 mg/dL and the upper limit of the laboratory normal range. The analysis of primary endpoint was based on investigator prescribed data.
Time Frame: 8 Weeks
Population: Intent to Treat (ITT) population, which includes all randomized subjects who received at least 1 dose of study drug and had at least 1 post-baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NPSP558 - 25 µg Dose | NPSP558 - 50 µg Dose
Number analyzed (Participants) | 19 | 23
percentage of participants | 21.1 [6.1 to 45.6] | 26.1 [10.2 to 48.4]
Statistical Analysis 1: Comparison: NPSP558 - 25 µg Dose vs NPSP558 - 50 µg Dose; The null hypothesis corresponding to the primary efficacy endpoint is that the percentages of subjects who meet the endpoint criteria are the same for both dose arms. This sample size for this study was not based on the statistical considerations; Test type: Superiority or Other; p > 0.999, Fisher Exact — All hypothesis testings in this study were based on type I error of 0.05. Adjustment for multiplicity was not applied; The 2-sided Fisher's Exact test was utilized to test for difference between the two dose arms; Treatment difference = 5.0, 95% CI 2-sided [-20.6 to 30.7] — The 2-sided asymptotic 95% confidence interval is based on normal approximation

2. Secondary Outcome: The Percentage of Subjects Who Met the Triple Efficacy Endpoint Criteria at Week 8.
Description: The triple efficacy endpoint criteria were defined as at least a 50% reduction from the baseline in oral calcium dose and at least a 50% reduction from the baseline in active vitamin D dose and an albumin-corrected total serum calcium concentration that was maintained or normalized compared to the baseline value (≥ 7.5 mg/dL) and did not exceed the upper limit of the laboratory normal range. The analysis of primary efficacy endpoint was based on investigator prescribed data
Time Frame: 8 Weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NPSP558 - 25 µg Dose | NPSP558 - 50 µg Dose
Number analyzed (Participants) | 19 | 23
percentage of participants | 10.5 [1.3 to 33.1] | 26.1 [10.2 to 48.4]
Statistical Analysis 1: Comparison: NPSP558 - 25 µg Dose vs NPSP558 - 50 µg Dose; The null hypothesis corresponding to this endpoint is that the percentages of subjects who meet the endpoint criteria are the same for both dose arms; Test type: Superiority or Other; p = 0.258, Fisher Exact; The 2-sided Fisher's Exact test was utilized to test for difference betweenthe two dose arms

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: 8 weeks on treatment
Arm/Group | NPSP558 - 25 µg Dose | NPSP558 - 50 µg Dose
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/23
Other Adverse Events (participants affected / at risk) | 11/19 | 17/23
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NPSP558 - 25 µg Dose (N=19) | NPSP558 - 50 µg Dose (N=23)
Paresthesia (Nervous system disorders) | 4 (8) | 5 (6)
Headache (Nervous system disorders) | 1 (1) | 3 (3)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (4)
Fatigue (General disorders) | 1 (1) | 2 (2)
Injection site pain (General disorders) | 0 (0) | 2 (4)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (5) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 2 (2)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other